CLINICAL TRIAL: NCT02608021
Title: Neurotrack Test Validation Protocol
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Neurotrack Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-00586
Record Dates: First submitted 2015-11-13; First posted 2015-11-18 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer's Disease; MRI
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amnestic mild cognitive impairment
- Cognitively normal

SUMMARY:
This protocol describes a study to validate Neurotrack's visual paired comparison task, aimed at early detection and monitoring of memory impairment. The investigators will determine whether the novel task developed by Neurotrack is associated with markers of brain pathology associated with very early Alzheimer's disease. The elderly subjects studied will be cognitively normal (CN) or have amnestic mild cognitive impairment (aMCI). For the current study, the primary brain pathology parameters will be derived from MRI scans. Data from this study will be correlated with data from a parallel study designed to validate a larger group of new cognitive tasks by correlating test performance with a broader array of biomarkers of Alzheimer's disease.

DETAILED DESCRIPTION:
The Neurotrack test has the potential to dramatically alter the current methods used for detecting cognitive deficits. Patients and research subjects could be screened for medial temporal lobe (MTL) impairment using inexpensive, widely available, safe, and non-invasive technology.

Subjects will be elderly individuals who are participating in ongoing research at the NYU Alzheimer's Disease Center (ADC) and who have received the standard ADC clinical evaluation within the past year, including a medical-neurological evaluation, neuro-psychological assessment and structural neuroimaging (MRI). As part of the current study, all subjects will receive both the Neurotrack Visual Paired-Comparison (VPC) Task and MRI scans. The current protocol strictly for a research study and there will be no "standard care" provided. Participants will be asked to come in for two separate sessions. The first session will involve screening to confirm eligibility and administration of the cognitive testing procedures, while the second session will involve the MRI protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis based on recent (within 1 year) consensus meeting, cross-referenced with standard neuropsychological scores:

   * Cognitively Normal (CN) Subjects: based on MMSE scores, CDR, and GDS.
   * Amnestic Mild Cognitive Impairment (aMCI) Subjects: Diagnosis of aMCI, based on MMSE scores, CDR, and GDS.
2. Normal or corrected-to-normal vision and hearing (able to see images on computer screen and hear auditory events delivered through the computer speaker).

Exclusion Criteria:

1. Significant history of mental illness, drug or alcohol abuse; severe trauma preventing normal use of dominant hand (needed to move the mouse cursor); clinical depression (unless medically controlled); other neurologic conditions (i.e. stroke), or learning disability; ophthalmologic/visual problems that prevent viewing a computer screen at a normal distance (such as legal blindness, detached retinas, occlusive cataracts).
2. Having pacemakers, aneurysm clips, cochlear implants, pulse oximeters, EKG leads, tattoos or other metal/foreign objects in body or face and therefore unable to receive MRI.
3. Lack the capacity to give informed consent and lack of an authorized surrogate to provide consent if the prospective subject is found to lack adequate consent capacity.
4. Pregnancy, breastfeeding or planning to have a baby.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals will be recruited from among participants at the NYU Alzheimer's Disease Center ADC, at the affiliated Center for Brain Health (CBH), and from other ongoing NYU research studies of the Center for Cognitive Neurology (CCN) that are affiliated with the ADC and for which participants receive the standard ADC research diagnostic assessment (the ADC Clinical Evaluation).
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Presence of eye fixation assessed by a point of gaze continually remaining within 1 degree of visual angle for a period of 100 milliseconds or more. | 2 months
  Eye fixation is defined as a point of gaze continually remaining within 1 degree of visual angle for a period of 100 milliseconds or more. Investigators will analyze the fixations that occur within 2 designated areas of interest (AOIs): the area of the novel image and the area of the familiar image.
Eye tracking data - Total looking time | 2 months
  Total looking time (i.e. the total sum of the duration for all fixations)
Eye tracking data - Total number of fixations | 2 months
  Total number of fixations (i.e. the total number of fixations that met the ≥100 ms criterion)
Eye tracking data - Percentage looking time | 2 months
  Percentage looking time on novel image

SECONDARY OUTCOMES:
Correlation of MRI data with VPC task score | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Ferris, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States